CLINICAL TRIAL: NCT06727266
Title: Ultrasonographic Evaluation of the Shoulder Joint in Patients With Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Berke Demir, doctor, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH-FTR-BD-001
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; ultrasonography; shoulder
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Axial Spondyloarthritis Patients: Demographic information such as age, height, weight and body mass index (BMI) will be recorded. During the physical examination, shoulder range of motion is measured and recorded. Shoulder pain will be assessed using the Visual Analogue Scale (VAS) and the Shoulder Pain and Disability Index (SPADI). Disease activity will be assessed using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). Functional status will be assessed using the Bath Ankylosing Spondylitis Functional Index (BASFI). Spinal mobility will be assessed using the Bath Ankylosing Spondylitis Metrology Index (BASMI). Shoulder imaging will be performed using a Mindray DC-8 ultrasound device in accordance with European Society of Musculoskeletal Radiology (ESSR) protocols.
  Interventions: Diagnostic Test: Shoulder ultrasound
- Healthy individuals: Demographic information such as age, height, weight and body mass index (BMI) will be recorded. During the physical examination, shoulder range of motion is measured and recorded. Shoulder pain will be assessed using VAS (Visual Analogue Scale) and SPADI (Shoulder Pain and Disability Index). Imaging of the shoulder joints will be performed using a Mindray DC-8 ultrasound machine according to European Society of Musculoskeletal Radiology (ESSR) protocols.
  Interventions: Diagnostic Test: Shoulder ultrasound

INTERVENTIONS:
Diagnostic Test: Shoulder ultrasound — The ultrasound examination is performed according to the protocols of the European Society of Musculoskeletal Radiology (ESSR). The tendons of the muscles forming the rotator cuff, the enthesis regions, the tendon of the long head of the biceps muscle, the subacromial-subdeltoid bursa, the acromioclavicular and glenohumeral joints are examined.

SUMMARY:
The aim of this observational study is to assess shoulder joint involvement in patients with axial spondyloarthritis using ultrasound and to compare the findings with those of healthy controls.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axial SpA) is a chronic inflammatory rheumatic disease that causes inflammation of the spine and sacroiliac joints. The condition usually begins at a young age (between 20 and 40 years). Common complaints include back pain, morning stiffness, and gradual restriction of spinal movement. Complaints of peripheral joint involvement may also be observed.

Shoulder involvement in patients with axial spondyloarthritis (axial SpA) represents a manifestation of the disease that can affect peripheral joints. Shoulder involvement typically develops as a result of an inflammatory process and is manifested by symptoms such as pain, swelling, and limitation of movement. The glenohumeral joint, acromioclavicular joint, subacromial bursa, and rotator cuff tendons are most commonly affected. Such peripheral joint involvement may indicate a more severe progression of axial SpA and an increased future disease burden.

Ultrasound is an inexpensive, non-invasive, and radiation-free imaging modality that is widely used in the assessment of the musculoskeletal system. In inflammatory rheumatic diseases such as axial SpA, ultrasound is a highly effective method for the early detection of inflammation. Inflammatory findings such as synovitis, tenosynovitis, enthesitis, and bursitis can be identified by ultrasound in the early stages of the disease. Early detection of these findings can slow disease progression and prevent joint damage by facilitating timely initiation of treatment.

The objective of this observational study is to evaluate the shoulder joint using ultrasound in patients with axial spondyloarthritis and to compare the findings with healthy controls.

The case group will consist of patients aged 18 to 65 who have been diagnosed with axial spondyloarthritis by a specialist in physical medicine and rehabilitation and who are being followed up at the PMR Outpatient Clinics of the Department of Physical Medicine and Rehabilitation, University of Health Sciences Gaziosmanpaşa Training and Research Hospital.

The control group will consist of individuals meeting the inclusion criteria, matched to the case group in terms of age and gender, and admitted to the PMR Outpatient Clinics of the Department of Physical Medicine and Rehabilitation, University of Health Sciences Gaziosmanpaşa Training and Research Hospital for any reason.

Physical examinations and ultrasound scans of the shoulder joint will be performed on all participants.

At the end of the study, data from both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a radiographic or non-radiographic diagnosis of axial spondyloarthritis according to ASAS 2009 classification criteria
* Patients aged 18-65
* For healthy controls; people aged 18-65 years who attended PMR outpatient clinics for any reason, without a diagnosis of inflammatory disease and without complaints of shoulder pain.

Exclusion Criteria:

* People under 18 and over 65
* History of shoulder trauma
* History of upper extremity surgery
* History of fracture of the upper extremity
* History of malignancy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Axial SpA patients and healthy volunteers (have close demographic data with Axial SpA patients)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Shoulder ultrasound findings | baseline
  Pathologies detected in the shoulder joint will be evaluated; tendon damage, bursitis, joint effusion, enthesitis etc.
  Enthesitis: Abnormal hypoechoic structure (loss of fibrillar structure of the tendon), thickening at the site of attachment of the tendon or ligament to the bone with associated Doppler signal and bone irregularities (calcification, cortical irregularity, enthesophyte).
  Synovitis: An abnormal hypoechoic intra-articular structure that is less compressed and may give a Doppler signal.
  Bursitis: Normally the bursa contains a thin layer of fluid, but in bursitis the amount of fluid increases and the bursa enlarges. There may be a marked thickening of the bursa walls. In bursitis, especially if it is chronic, septations (membrane formations) may be seen within the bursa.
  Effusion: Increased fluid in the joint space, manifested as anechoic fluid.
  Erosion: Causes irregularity or disruption of the normally flat bone cortex.

SECONDARY OUTCOMES:
BASDAI | baseline
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): It consists of six questions about five main symptoms, including fatigue, spinal pain, joint pain or swelling, localised tenderness and morning stiffness.The final BASDAI score ranges from 0 to 10, and higher scores represent higher disease activity.
BASFI | baseline
  Bath Ankylosing Spondylitis Functional Index (BASFI): BASFI is an easy-to-administer, sensitive and reliable self-report questionnaire developed to assess physical function in AS patients. It consists of a total of 10 items. The BASFI Score is the average of the 10 items and ranges from 0 to 10, with higher scores indicating more functional limitations.
BASMI | baseline
  Bath Ankylosing Spondylitis Metrology Index (BASMI): It is an index consisting of tragus wall, cervical rotations, lumbar lateral flexions, modified Schober and intermalleolar distance measurements.
VAS | baseline
  A 100 mm line is drawn, and the two ends of the line are labeled with the two extreme descriptions of pain. The patient is asked to mark their current level of pain on this line. One end of the line is labeled "no pain," and the other end is labeled "severe pain." The patient marks their current condition on the line. The distance from the "no pain" point to where the patient marks on the line represents the intensity of the patient's pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Research and Education Hospital, Istanbul, Turkey (Türkiye)